CLINICAL TRIAL: NCT00246532
Title: Opiate-Induced Tolerance & Hyperalgesia in Pain Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Dr. Lawrence Chu, National Institute of General Medical Sciences, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 5K23GM071400-02 (NIH); 5K23GM071400-02 (NIH)
Record Dates: First submitted 2005-10-26; First posted 2005-10-31 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Chronic Low Back Pain; Opioid-induced Hyperalgesia
MeSH Terms: interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1: Placebo Pill (Placebo Comparator): This arm contains placebo medication.
  Interventions: Drug: Placebo
- 2: Morphine (Active Comparator): Patients will receive oral morphine therapy.
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Morphine — Patients will be given morphine sulfate oral medication until their back pain is adequately controlled.
  Arms: 2: Morphine
Drug: Placebo — Patients will receive placebo tablets.
  Arms: 1: Placebo Pill

SUMMARY:
Opiates such as morphine are the cornerstone medications for the treatment of moderate to severe pain. Recent evidence suggests that pain patients on chronic opioid therapy become more sensitive to pain (hyperalgesia) over time. There is also a long-standing notion that analgesic tolerance to opioids (habituation) develops during chronic use even though this phenomenon has never been prospectively studied. Our specific aims propose to prospectively test the hypotheses that; 1) Pain patients on chronic opioid therapy develop dose-dependent tolerance and/or hyperalgesia to these medications over time, 2) Opioid-induced tolerance and hyperalgesia develop differently with respect to various types of pain, 3) Opioid-induced hyperalgesia occurs independently of withdrawal phenomena, and 4) Opioid-induced tolerance and hyperalgesia develop differently based on gender and/or ethnicity. This proposed study will be the first quantitative and prospective study of tolerance and hyperalgesia in pain patients and will have important implications for the rational use of opioids in the treatment of chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* opioid naïve (or less than 4 vicodin equiv/day)
* 18-70 years old
* candidate for opioid therapy for nonmalignant pain.

Exclusion Criteria:

* history of substance abuse or severe psychiatric disease
* use of medications for the treatment of neuropathic pain as these may alter tolerance or hyperalgesia
* neurological conditions interfering with experimental pain testing, e.g. severe peripheral neuropathy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2005-10; Primary Completion 2008-12 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Pain Tolerance | 1 month
Pain Threshold | 1 month

SECONDARY OUTCOMES:
Opioid Titration | 1 month
Pain Intensity | 1 month
Roland-Morris Disability Index | 1 month
Beck Depression Inventory | 1 month
Follow-Up Survey | 1 year
  Patients were asked about their average pain levels and current medication usage

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence F Chu, MD, MS, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States